CLINICAL TRIAL: NCT04030533
Title: A Study to Evaluate the Pharmacokinetics of Guselkumab and Ustekinumab Following a Single Intravenous or Subcutaneous Administration in Healthy Chinese Subjects
Brief Title: Study of Guselkumab and Ustekinumab Following a Single Intravenous or Subcutaneous Administration in Healthy Chinese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: CR108639; CNTO1959CRD1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2019-07-22; First posted 2019-07-24 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — guselkumab; Ustekinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Cohort 1: Guselkumab (SC): Dose 1 (Experimental): Participants will receive a single subcutaneous (SC) injection of guselkumab (dose 1), administered on Day 1.
  Interventions: Drug: Guselkumab (SC): Dose 1
- Cohort 2: Guselkumab (SC): Dose 2 (Experimental): Participants will receive a single SC injection of guselkumab (dose 2), administered on Day 1.
  Interventions: Drug: Guselkumab (SC): Dose 2
- Cohort 3: Guselkumab (IV): Dose 1 (Experimental): Participants will receive a single intravenous (IV) infusion of guselkumab (dose 1), administered on Day 1.
  Interventions: Drug: Guselkumab (IV): Dose 1
- Cohort 4: Guselkumab (IV): Dose 2 (Experimental): Participants will receive a single IV infusion of guselkumab (dose 2), administered on Day 1.
  Interventions: Drug: Guselkumab (IV): Dose 2
- Cohort 5: Ustekinumab (IV): 6 mg/mL (Experimental): Participants will receive a single IV infusion of ustekinumab 6 milligrams per milliliter (mg/mL) solution on Day 1.
  Interventions: Drug: Ustekinumab 6 mg/mL

INTERVENTIONS:
Drug: Guselkumab (SC): Dose 1 — Participants will receive a single dose of guselkumab (dose 1) subcutaneously.
  Other Names: CNTO 1959
  Arms: Cohort 1: Guselkumab (SC): Dose 1
Drug: Guselkumab (SC): Dose 2 — Participants will receive a single dose of guselkumab (dose 2) subcutaneously.
  Other Names: CNTO 1959
  Arms: Cohort 2: Guselkumab (SC): Dose 2
Drug: Guselkumab (IV): Dose 1 — Participants will receive a single IV infusion of guselkumab (dose 1).
  Other Names: CNTO 1959
  Arms: Cohort 3: Guselkumab (IV): Dose 1
Drug: Guselkumab (IV): Dose 2 — Participants will receive a single IV infusion of guselkumab (dose 2).
  Other Names: CNTO 1959
  Arms: Cohort 4: Guselkumab (IV): Dose 2
Drug: Ustekinumab 6 mg/mL — Participants will receive a single IV infusion of ustekinumab 6 mg/mL solution.
  Other Names: Stelara
  Arms: Cohort 5: Ustekinumab (IV): 6 mg/mL

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (PK) of guselkumab following a single intravenous (IV) or subcutaneous (SC) administration in healthy Chinese participants; to evaluate the PK of ustekinumab following a single IV administration in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be healthy with no clinically significant abnormalities as determined by medical history, physical examination, blood chemistry assessments, hematologic assessments, urinalysis, measurement of vital signs, and electrocardiogram (ECG)
* A woman must have a negative highly sensitive serum (beta-human chorionic gonadotropin [beta-hCG]) at screening and Day-1
* Must agree to use an adequate contraception method as deemed appropriate by the investigator; to always use a condom during intercourse and to not donate sperm during the study and for 16 weeks after study drug administration
* Must be a nonsmoker or agree to smoke no more than 10 cigarettes or 2 cigars per day throughout the study. However, during the inpatient portion of the study if smoking is not allowed in the inpatient unit, smokers will not be allowed to smoke cannot use nicotine replacement products
* Must agree to abstain from alcohol intake 48 hours before study drug administration and during the inpatient period of the study. After this time, participants must not consume more than 10 grams of alcohol (e.g. 250 milliliter (mL) beer with 5 percent (%) alcohol content) per day for the duration of the study

Exclusion Criteria:

* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, neurologic or psychiatric disease, infection, gastro-intestinal disease, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Has had major surgery, (for example, requiring general anesthesia) within 12 weeks before screening, or will not have fully recovered from surgery, or has surgery planned during the time the participant is expected to participate in the study
* Has known allergies, hypersensitivity, or intolerance to guselkumab or its excipients
* Has received an experimental antibody or biologic therapy within the previous 6 months
* Has a history of, or ongoing, chronic, or recurrent infectious disease, including but not limited to, chronic renal infection, chronic chest infection, recurrent urinary tract infection

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-11-29 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) | Predose (Day 1), 1, 4, 12, 24, 48, 72, 96, 120, and 144 hours postdose (Day 7); Days 15, 22, 29, 43, 57, 71, and 85
  The Cmax is the maximum observed serum concentration.
Area Under the Serum Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) | Predose (Day 1), 1, 4, 12, 24, 48, 72, 96, 120, and 144 hours postdose (Day 7); Days 15, 22, 29, 43, 57, 71, and 85
  AUC (0-infinity) is the area under the serum concentration versus time curve from time zero to infinity with extrapolation of the terminal phase.
Area Under Serum Concentration From Time Zero to the Last Quantifiable Concentration (AUC [0-last]) | Predose (Day 1), 1, 4, 12, 24, 48, 72, 96, 120, and 144 hours postdose (Day 7); Days 15, 22, 29, 43, 57, 71, and 85
  AUC (0-last) area under the serum concentration versus time curve from time zero to the time corresponding to the last quantifiable concentration.
Elimination Half-Life (T1/2) | Predose (Day 1), 1, 4, 12, 24, 48, 72, 96, 120, and 144 hours postdose (Day 7); Days 15, 22, 29, 43, 57, 71, and 85
  Elimination half-life is time measured for the serum concentration to decrease by 1 half to its original concentration. It is associated with the terminal slope of the semi logarithmic drug concentration-time curve, and is calculated as 0.693/lambda(z).
Total Systemic Clearance (CL) | Predose (Day 1), 1, 4, 12, 24, 48, 72, 96, 120, and 144 hours postdose (Day 7); Days 15, 22, 29, 43, 57, 71, and 85
  CL is a quantitative measure of the rate at which a drug substance is removed from the body. The total systemic clearance after intravenous dose is estimated by dividing the total administered dose by the serum area under the serum concentration-time curve from time zero to infinite time (AUC [0-infinity]).
Volume of Distribution (Vz) | Predose (Day 1), 1, 4, 12, 24, 48, 72, 96, 120, and 144 hours postdose (Day 7); Days 15, 22, 29, 43, 57, 71, and 85
  The Vz is total volume of distribution at terminal phase after intravenous (IV) administration, defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug.
Time to Reach Maximum Observed Serum Concentration (Tmax) | Predose (Day 1), 1, 4, 12, 24, 48, 72, 96, 120, and 144 hours postdose (Day 7); Days 15, 22, 29, 43, 57, 71, and 85
  Tmax is time correspondent to the maximum observed serum concentration.
Apparent Total Systemic Clearance (CL/F) | Predose (Day 1), 1, 4, 12, 24, 48, 72, 96, 120, and 144 hours postdose (Day 7); Days 15, 22, 29, 43, 57, 71, and 85
  Apparent total systemic clearance is clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Apparent Volume of Distribution (Vz/F) | Predose (Day 1), 1, 4, 12, 24, 48, 72, 96, 120, and 144 hours postdose (Day 7); Days 15, 22, 29, 43, 57, 71, and 85
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired serum concentration of a drug. Apparent volume of distribution after subcutaneous dose (Vz/F) is influenced by the fraction absorbed.
Absolute Bioavailability (F [%]) | Predose (Day 1), 1, 4, 12, 24, 48, 72, 96, 120, and 144 hours postdose (Day 7); Days 15, 22, 29, 43, 57, 71, and 85
  Absolute bioavailability is the percentage of the orally administered dose that is systemically available. It is calculated as (AUC [0-infinity] for test)/(AUC [0-infinity] for reference [ref])*(D for ref/D for test)*100, where the reference treatment is an intravenous administration, AUC (0-infinity) is area under the concentration-time curve from time zero to extrapolated infinite time, and D is the dose of administered drug.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Up to Week 16
  An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Number of Participants with Anti-Guselkumab and Anti-Ustekinumab Antibodies | Predose (Day 1) and on Days 15, 29, 57, and 85
  Participant's serum samples will be collected and screened for antibodies binding to guselkumab and ustekinumab using validated electrochemiluminescence immunoassay analyzer (ECLIA) method for evaluation of potential immunogenicity.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency